CLINICAL TRIAL: NCT00134771
Title: Trial of Nutritional Supplementation in Infants Born Small for Gestational Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 99/2/109
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2005-08

CONDITIONS: Birth Weight
Keywords: Infants whose birthweight is less than the 20th centile for gestational age (UK standards); Infants who are formula fed from birth; Singletons; Infants free from major congenital disease
MeSH Terms: conditions — Birth Weight

INTERVENTIONS:
Drug: Nutrient enriched infant formula

SUMMARY:
The purpose of this study was to determine whether giving a nutrient enriched formula to infants born small-for-gestational age benefits blood pressure, growth and body composition by six months of age.

DETAILED DESCRIPTION:
Infants born small for gestational age often show impaired growth during childhood and reduced height as adults. Infants who are breast-fed from birth show greater 'catch-up' growth during the first few months of life than those who are formula fed but it is not clear what factors in breast milk (ie protein, nucleotides, LCPUFAs) are responsible for this 'catch-up' growth. This RCT compares the effects of using an enriched formula with increased protein and modified triglyceride (palmitate predominantly in Sn-2 position) against a standard infant formula from birth to six months on infants whose birth weights are below the 20th centiles for gestational age.

Infants are measured by a research midwife within 10 days of birth (at randomisation), 8, 16 and 26 weeks of age. At randomisation consent from the mother is taken and information collected about the pregnancy, social, demographic and medical data. At this and each further visit anthropometric measurements including skinfolds will be collected in addition to blood pressure and bio-electrical impedence at six months. A sub-sample of infants will have their body composition assessed by deuterium labelled water at six months. Data on health, weaning diets and bowel function are also collected at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are formula fed from birth
* Infants whose birthweights are less than 20th centile
* Singleton births
* Gestation > 37 weeks
* Infants free from major congenital disease

Exclusion Criteria:

* Infants who are breast-fed
* Multiple births
* Birthweight > 20th centile
* Infants with congenital disease
* Gestation < 37 weeks

Ages: 0 Years to 10 Days | Sex: All
Age Groups: Child
Dates: Start 2001-02; Study Completion 2003-06

PRIMARY OUTCOMES:
Weight, length, head circumference at 6 months

SECONDARY OUTCOMES:
Body composition at 6 months
Blood pressure at six months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Singhal, Principal Investigator — Institute of Child Health
Locations (6):
- United Kingdom (6):
  - Neonatal Unit, Wishaw Hospital, 50 Netherton St, Wishaw, Lanrkshire
  - The Queen Mother's Hospital, Yorkhill, Glasgow
  - Maternity Hospital, Glasgow Royal Infirmary, Glasgow
  - Maternity Unit, Southern General Hospital, 1345 Govan Road, Glasgow
  - MRC Childhood Nutrition Research Centre, Inst of Child Health, London
  - Maternity Unit, Royal Alexandra Hospital, Corsebar Road, Paisley